CLINICAL TRIAL: NCT05065411
Title: P3 Efficacy Evaluation of Enobosarm in Combo With Abemaciclib Compared to Estrogen Blocking Agent for 2nd Line Treatment of ER+HER2- MBC in Patients Who Have Shown Previous Disease Progression on an Estrogen Blocking Agent Plus Palbociclib
Brief Title: Efficacy & Safety Evaluation of Enobosarm in Combo With Abemaciclib in Treatment of ER+HER2- Metastatic Breast Cancer
Acronym: VERU-024
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Veru Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V2000701
Record Dates: First submitted 2021-09-21; First posted 2021-10-04 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ostarine; abemaciclib; exemestane; Everolimus; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Open Label two treatment arm
Who Masked: Outcomes Assessor
Masking Description: Only the central radiologist readers will be blinded to treatment assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enobosarm Combination Group (Experimental): Enobosarm Combination Group will receive enobosarm 9 mg each day by mouth (QD), and abemaciclib will administered by mouth at a dose of 150 mg BID.
  Stage 2 Subjects in the Enobosarm Combination Group will receive enobosarm 9 mg QD each day by mouth and abemaciclib 150 mg BID by mouth until disease progression is observed and confirmed by BICR.
  Interventions: Drug: Enobosarm & Abemaciclib Combo
- Control Treatment Group (Active Comparator): Control Treatment Group will receive a non-steroidal AI, a non-steroidal or steroidal (exemestane with or without everolimus), AI OR fulvestrant approved for the treatment of metastatic breast cancer and is part of the standard of care at the clinical study site until disease progression is observed and confirmed by BICR. The decision of which comparator treatment will be used will be made prior to randomization.
  Interventions: Drug: non-steroidal AI, or steroidal AI (exemestane with or without everolimus) or Fulvestrant

INTERVENTIONS:
Drug: Enobosarm & Abemaciclib Combo — Subjects will receive a combo of Enobosarm & Abemaciclib
  Other Names: VERU-024; Verzenio
  Arms: Enobosarm Combination Group
Drug: non-steroidal AI, or steroidal AI (exemestane with or without everolimus) or Fulvestrant — Non-steroidal AI, a steroidal AI (exemestane with or without everolimus), OR fulvestrant
  Other Names: exemestane; fulvestrant; exemestane plus everolimus
  Arms: Control Treatment Group

SUMMARY:
STAGE 1: To determine the safety of enobosarm 9 milligram (mg) once daily (QD) used in combination with a CDK 4/6 inhibitor [Verzenio® (abemaciclib) tablets, for oral use, 150 mg twice daily (BID)].

STAGE 2: To demonstrate the efficacy and safety of enobosarm 9 mg QD in combination with abemaciclib 150 mg BID (Enobosarm Combination Group) versus Estrogen Blocking Agent (Control Treatment Group) in the treatment of estrogen receptor positive (ER+), human epidermal growth factor receptor 2 negative (HER2-), androgen receptor positive (AR+) with a AR% nuclei staining ≥40% metastatic breast cancer that have previously experienced disease progression on an estrogen blocking agent plus (palbociclib) as measured by progression free survival (PFS) according to RECIST 1.1 criteria.

DETAILED DESCRIPTION:
STAGE 1: This is an open-label safety study of enobosarm 9 mg QD coadministered with a CDK 4/6 inhibitor (abemaciclib), 150 mg BID.

STAGE 2: This study is a multicenter, randomized, open-label, two treatment arm, efficacy and safety study. Subjects will be randomized to the two treatment arms (Enobosarm Combination Group versus Control Treatment Group) in a 1:1 fashion. The determination of the treatment to be used in the control arm will be declared prior to randomization.

If first line of therapy for metastatic breast cancer was a non-steroidal AI plus palbociclib, then the patient will be randomized to either enobosarm + abemaciclib OR fulvestrant.

If first line of therapy for metastatic breast cancer was fulvestrant plus palbociclib, then the patient will be randomized to either enobosarm + abemaciclib OR AI (steroidal or non-steroidal). If the patient is randomized to the Control Treatment Group to receive steroidal AI, (exemestane) the patient may receive exemestane with or without everolimus.

The primary efficacy endpoint of the study will be the median PFS as defined by RECIST 1.1.

Subjects will continue study treatment until disease progression confirmed by blinded independent central reader (BICR) is observed. A safety follow up visit will occur approximately 30 days after last dose of study drug.

Long term survival follow up - every 30 days after last dose of study drug for 1 year and then every 90 days thereafter.

ELIGIBILITY:
Inclusion Criteria:

Subjects accepted for this study must:

* Provide informed consent
* Be able to communicate effectively with the study personnel
* Aged ≥18 years
* For Female Subjects

  * Menopausal status
  * Be postmenopausal as defined by the National Comprehensive Cancer Network as either: Age ≥55 years and one year or more of amenorrhea Age <55 years and one year or more of amenorrhea, with an estradiol assay <20 pg/mL Age <55 years and surgical menopause with bilateral oophorectomy
  * Be premenopausal or perimenopausal with a negative serum pregnancy test.
  * If subject is of child bearing potential, the subject must agree to use acceptable methods of contraception:
* If female study participant could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 6 months following administration of the last dose of study medication. Acceptable methods of contraception are as follows: Condom with spermicidal foam/gel/film/cream/suppository [i.e., barrier method of contraception], surgical sterilization of male partner (vasectomy with documentation of azoospermia) and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository},
* If female study participant has undergone documented tubal ligation (female sterilization), a barrier method (condom used with spermicidal foam/gel/film/cream/suppository) should also be used
* If female study participant has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS), a barrier method (condom with spermicidal foam/gel/film/cream/suppository) should also be used
* For Male Subjects

Subject must agree to use acceptable methods of contraception:

* If the study subject's partner could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 6 months following administration of the last dose of study medication. Acceptable methods of contraception are as follows: Condom with spermicidal foam/gel/film/cream/suppository [i.e., barrier method of contraception], surgical sterilization (vasectomy with documentation of azoospermia) and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository}, the female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method (condom used with spermicidal foam/gel/film/cream/suppository)
* If female partner of a study subject has undergone documented tubal ligation (female sterilization), a barrier method (condom used with spermicidal foam/gel/film/cream/suppository) should also be used
* If female partner of a study subject has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS), a barrier method (condom with spermicidal foam/gel/film/cream/suppository) should also be used

  * For premenopausal and perimenopausal women where exemestane monotherapy or exemestane plus everolimus is chosen as the active control treatment patient must be already on ovarian suppression or to be candidates for this treatment: e.g., luteinizing hormone release hormone agonist or ovariectomy
  * Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
  * Documented evidence of ER+HER2- metastatic breast cancer (NOTE: patients with HER2+ metastatic breast cancer are excluded from participation in this study)
  * Measurable disease is required as per RECIST 1.1 (NOTE: Bone only metastatic disease is acceptable but requires a measurable component)
  * Have AR% nuclei staining ≥40% as assessed by central laboratory
  * Previously treated (and progressed on) with the following:

    * nonsteroidal aromatase inhibitor plus palbociclib for metastatic breast cancer OR
    * fulvestrant plus palbociclib for metastatic breast cancer
  * Subject is willing to comply with the requirements of the protocol through the end of the study
  * Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and randomization.
  * Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization
  * The patient is able to swallow oral medications
  * The patient has adequate organ function for all of the following criteria, as defined in Table 1 of the Protocol

Exclusion Criteria:

Any of the following conditions are cause for exclusion from the study:

* Known hypersensitivity or allergy to enobosarm or abemaciclib
* Patients with a biliary catheter
* Creatinine clearance < 30 milliliter per minute (mL/min) as measured using the Cockcoft Gault formula (patients with mild and moderate renal failure are not excluded from participation in this study)
* Previously received >1 course of systemic chemotherapy (not including immunotherapies or targeted therapies) for the treatment of metastatic breast cancer.

NOTE: Subjects may have received 1 course of chemotherapy in the adjuvant or neoadjuvant setting would not count as a line of therapy.

* Subjects with radiographic evidence of central nervous system (CNS) metastases as assessed by CT or MRI that are not well-controlled (symptomatic or requiring control with continuous corticosteroid therapy [e.g., dexamethasone]) NOTE: Subjects with CNS metastases are permitted to participate in the study if the CNS metastases are medically well-controlled and stable for at least 30 days after receiving local therapy (irradiation, surgery, etc.)
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Treatment with any investigational product within < 4 half-lives for each individual investigational product OR within 30 days prior to randomization
* Major surgery within 30 days prior to randomization
* Testosterone, methyltestosterone, oxandrolone (Oxandrin®), oxymetholone, danazol, fluoxymesterone (Halotestin®), testosterone-like agents (such as dehydroepiandrosterone, androstenedione, and other androgenic compounds, including herbals), or antiandrogens (flutamide, bicalutamide, abiraterone, enzalutamide, apalutamide, or darolutamide). Previous therapy with testosterone and testosterone-like agents is acceptable with a 30-day washout (if previous testosterone therapy was long term depot within the past 6 months, the site should contact the Medical Monitor) or any other androgenic agent.
* Treatment with any of the following hormone therapies for metastatic breast cancer. Prior use in the adjuvant or neoadjuvant setting is allowed if the treatment is discontinued greater than 30 days prior to randomization

  * Estrogens
  * Megestrol acetate
  * Testosterone
* All other concurrent anticancer treatments (including, but not limited to, all SERMs, estrogen blocking agents unless randomized to Control Treatment Group, and CDK 4/6 inhibitors unless randomized to the abemaciclib in Enobosarm Combination Group)
* An abnormal ECG result which, based on the investigator's clinical judgment, would place the subject at increased risk
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Has a known additional, invasive, malignancy that is progressing or required active treatment in the last 5 years [note: subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, ductal breast carcinoma in situ, bladder cancer (superficial curatively treated), or cervical carcinoma in situ that have undergone potentially curative therapy are not excluded]
* Pregnant, lactating, or breastfeeding, or intending to become pregnant during the study or within 60 days after the final dose of study treatment
* The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Primary endpoint for the study is the median progression free survival (PFS) in the Enobosarm Combination Group compared to the Control Treatment Group in patients with AR% nuclei staining ≥40%. Progression will be defined based on RECIST 1.1 criteria | Day 1 to Day 300
  STAGE 1: To determine the safety of enobosarm 9 mg once daily (QD) used in combination with abemaciclib tablets, for oral use, 150 mg twice daily (BID)].
  STAGE 2: To demonstrate the efficacy of enobosarm in combination with abemaciclib (Enobosarm Combination Group) versus an estrogen blocking agent, (non-steroidal AI, steroidal AI (exemestane with or without everolimus) or fulvestrant Control Treatment Group) in the treatment of AR+ER+HER2 (AR% nuclei staining ≥40%) metastatic breast cancer as measured by PFS according to RECIST 1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR), proportion of subjects with a best tumor response of ORR (partial response [PR] or complete response [CR]) on study | Day 1 to Day 300
  Objective Response Rate (ORR), proportion of subjects with a best tumor response of ORR (partial response [PR] or complete response [CR]) on study

CONTACTS AND LOCATIONS:
Overall Officials: Barnette, Study Chair — Veru Inc.
Locations (30):
- United States (30):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Banner MDACC, Gilbert, Arizona
  - Arizona Oncology Associates, PC-HOPE, Tucson, Arizona
  - Los Angeles Cancer Network One Oncology, Los Angeles, California
  - UCLA Parkside Cancer Center, Los Angeles, California
  - Sharp Center for Research, San Diego, California
  - Sansum Clinic, CA, Santa Barbara, California
  - Innovative Clinical Research Institute, Whittier, California
  - Med OncologyHematology Consultants, PA Newark, Newark, Delaware
  - Lakes Research, Miami Lakes, Florida
  - Maryland Oncology Hematology, P.A., Annapolis, Maryland
  - Baystate Regional Cancer Program - D'Amour Center for Cancer Care, Springfield, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University St. Louis, St Louis, Missouri
  - Renown Health, Reno, Nevada
  - Summit Medical Group, Florham Park Campus, Florham Park, New Jersey
  - The New York Hospital, Westbury, New York
  - The Lindner Center for Research and Education at the Christ Hospital, Cincinnati, Ohio
  - Toledo Clinic Cancer Centers - Main Office, Toledo, Ohio
  - UPMC Magee-Women's Hospital, Pittsburgh, Pennsylvania
  - Texas Oncology, PA, Dallas, Texas
  - Texas Oncology, PA, Denton, Texas
  - Texas Oncology, P.A., El Paso, Texas
  - Texas Oncology, P.A., Flower Mound, Texas
  - UT MD Anderson CC, Houston, Texas
  - Texas Oncology, P.A., San Antonio, Texas
  - Texas Oncology, P.A., Tyler, Texas
  - Virginia Oncology Assoc, Norfolk, Virginia
  - University of Washington Seattle Cancer Center Alliance (SCCA), Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided